CLINICAL TRIAL: NCT02481466
Title: The First Cross-Canada Trial of the Nutrition Trialists' Network--Enhanced Dietary Portfolio and Exercise on Arterial Damage (MRI-Enhanced Dietary Portfolio Plus Exercise on Cardiovascular Risk)
Brief Title: The Combined Portfolio Diet and Exercise Study
Acronym: PortfolioEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other); Laval University (Other); University of Manitoba (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: REB # 14-316; FRN 130278 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR)); FRN 129920 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2015-05-26; First posted 2015-06-25 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Diseases; Hypercholesterolemia; Type 2 Diabetes; Metabolic Syndrome
Keywords: Arterial plaque; Magnetic resonance imaging (MRI); Portfolio diet; Dietary modification; Dietary trials; hypercholesterolemia; diabetes; exercise; cardiovascular disease risk; glycemic index (GI); Carotid Ultrasound; Dietary Approaches to Stop Hypertension (DASH) diet
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia; Diabetes Mellitus, Type 2; Metabolic Syndrome; Diabetes Mellitus; Motor Activity | interventions — Diet

STUDY DESIGN:
Intervention Model Description: This is a 2 x 2 factorial design
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Portfolio diet and structured exercise (Experimental): Participants will receive advice on a therapeutic diet appropriate for hypercholesterolemia (ie <7% of energy from saturated fat, <200mg/d cholesterol) PLUS the combination of viscous fibres, soy protein, plant sterols and nuts, 5% extra monounsaturated fat, and selection of low glycemic index foods and be instructed on a standardized physical activity/exercise component supervised by kinesiologists.
  Interventions: Behavioral: Portfolio diet and structured exercise
- DASH-like diet and structured exercise (Active Comparator): Participants will receive advice to follow a DASH-like diet of whole grains, and low-fat dairy products with fruits and vegetables and a be instructed on the Laval exercise program-a standardized physical activity/exercise component supervised by trained kinesiologists (exercise physiologists).
  Interventions: Behavioral: DASH-like diet and structured exercise
- Portfolio diet and routine exercise (Experimental): Participants will receive advice that will conform to the current therapeutic diet appropriate for hypercholesterolemia (ie <7% of energy from saturated fat, <200mg/d cholesterol) PLUS the combination of viscous fibres, soy protein, plant sterols and nuts, 5% extra monounsaturated fat, and selection of low glycemic index foods and will be provided with a copy of Health Canada Physical Activity Guidelines with advice to increase physical activity.
  Interventions: Behavioral: Portfolio diet and routine exercise
- DASH-like diet and routine exercise (Active Comparator): Participants will receive advice to follow a DASH-like diet of whole grains, and low-fat dairy products with fruits and vegetables and will be provided with a copy of Health Canada Physical Activity Guidelines with advice to increase physical activity.
  Interventions: Behavioral: DASH-like diet and routine exercise

INTERVENTIONS:
Behavioral: Portfolio diet and structured exercise — Diet: Foods will contribute 9 g/1000 kcal viscous fibre as β-glucan (oats, barley and oat bran breads) and psyllium (cereal), 1 g plant sterol/1000 kcal diet (in sterol margarine), 22.5 g soy protein/1000 kcal (soy burgers and other soy meat analogues, soy milks, yogurts and cheese) and 22.5 g nuts/1000 kcal and increased MUFA (as olive and canola oils, avocados, nuts etc.). The glycemic index will be reduced from 83 to 70 GI units (bread scale).
  Exercise: A program encouraging 150 minutes of exercise, based on the Quebec Heart and Lung Institute exercise program. A short submaximal treadmill test will be used to assess cardiorespiratory fitness. A kinesiologist will work with participants using behavioral strategies to achieve the target of 150 min/week of physical activity or exercise in 3 or 5 sessions weekly (vigorous, moderate or mild depending on goals and tolerance). The target goal will be at least 10,000 steps daily.
  Other Names: Dietary Portfolio of cholesterol-lowering foods; Enhanced portfolio; Low Glycemic Index Portfolio; Portfolio Plus diet; Laval exercise program; structured exercise program; Portfolio diet; structured exercise
  Arms: Portfolio diet and structured exercise
Behavioral: DASH-like diet and structured exercise — Diet: Participants will be encouraged to follow a diet of whole grain foods (brown rice, whole wheat breads, muffins and breakfast cereals), reduce meat consumption, choose low fat dairy foods and a control margarine.
  Exercise: A physical activity/exercise program encouraging 150 minutes of exercise, based on the exercise program developed at the Quebec Heart and Lung Institute. A short submaximal treadmill test will be used to assess cardiorespiratory fitness. A kinesiologist will work with participants using behavioral strategies to develop and support a plan that aims to achieve the target of 150 min/week of physical activity or exercise in 3 or 5 sessions weekly (vigorous, moderate or mild depending of goals and tolerance) in keeping with maximum achievable goals of participants. The target goal will be at least 10,000 steps daily recorded on their pedometers.
  Other Names: Modified DASH diet; high fibre diet; structured exercise program; DASH-like diet; Laval exercise program
  Arms: DASH-like diet and structured exercise
Behavioral: Portfolio diet and routine exercise — Diet: Foods on the dietary portfolio plan will contribute 9 g/1000 kcal viscous fibre as β-glucan (oats, barley and oat bran breads) and psyllium (cereal), 1 g plant sterol/1000 kcal diet (in sterol margarine), 22.5 g soy protein/1000 kcal (soy burgers and other soy meat analogues, soy milks, yogurts and cheese) and 22.5 g peanuts or equivalent of tree nuts/1000 kcal (Table 1A) and increased MUFA (as olive and canola oils, avocados, nuts etc.). The glycemic index will be reduced from 83 to 70 GI units (bread scale).
  Exercise: Participants in this group will receive standard of care for individuals being seen by a general practitioner. They will be advised to achieve the current recommended targets for daily physical activity and educational material published by Health Canada (Canada's Physical Activity Guide, Health Canada). They will undergo treadmill tests at the start and end of each 1 year period. They will not receive the more frequent, targeted visits with a kinesiologist.
  Other Names: Dietary Portfolio of cholesterol-lowering foods; Enhanced portfolio; Low Glycemic Index Portfolio; Portfolio Plus diet; routine exercise
  Arms: Portfolio diet and routine exercise
Behavioral: DASH-like diet and routine exercise — Diet: Participants will be encouraged to follow a diet of whole grain foods (brown rice, whole wheat breads, muffins and breakfast cereals), reduce meat consumption, choose low fat dairy foods and a control margarine.
  Exercise: Participants in this group will receive standard of care for individuals being seen by a general practitioner. They will be advised to achieve the current recommended targets for daily physical activity and educational material published by Health Canada (Canada's Physical Activity Guide, Health Canada). They will undergo treadmill tests at the start and end of each 1 year period. They will not receive the more frequent, targeted visits with a kinesiologist.
  Other Names: Modified DASH diet; high fibre diet; routine exercise
  Arms: DASH-like diet and routine exercise

SUMMARY:
The purpose of this study is to determine whether a dietary portfolio of cholesterol-lowering foods (viscous fibres, soy protein, plant sterols and nuts) further enhanced by increased levels of monounsaturated fatty acids (MUFA) and low glycemic index foods; together with a structured exercise program reduce the progression of carotid and coronary atheromatous lesions, Low density lipoprotein-cholesterol (LDL-C), and blood pressure, while reducing the number of individuals requiring statins.

DETAILED DESCRIPTION:
Presently in Canada, 29% of deaths are due to cardiovascular disease (CVD), costing $20.9 billion annually. The investigators have, therefore, brought together an unique network of investigators at different stages in their careers with a range of disciplines (nutrition, cardiology, diabetes, exercise physiology, imaging, physics, clinical trials, statistics, laboratory medicine, primary care, genetics, psychology, knowledge translation (KT), epidemiology), and with international recognition, experience and connections, to undertake a Canada-wide, multi-centre study which will test the ability of an effective cholesterol-lowering diet (dietary portfolio) and an exercise program, developed at Laval University, over 3 years to reduce the progression of plaque build-up in the carotid artery as assessed by Magnetic Resonance Imaging (MRI) in individuals with hypercholesterolemia and or type 2 diabetes. The dietary portfolio which has been proven in many of our studies to be an effective cholesterol-lowering diet will be enhanced to include features from other dietary strategies which the investigators have tested or developed; such as high monounsaturated fat (from Mediterranean diet) (CMAJ 2010) and low glycemic index foods (JAMA 2008). The investigators plan to recruit194 (approximately 200) men and postmenopausal women, who have measurable thickening (as assessed by ultrasound) due to plaque build up in the carotid arteries, in a 1.5 year period for this 3 year study. Ultrasound selection will be of individuals with intima-media thickness (IMT) >/=1.2mm as relevant arterial thickening to ensure a relatively low risk for the majority of the group, yet with some measurable arterial thickening.

Those selected will be randomly assigned to receive advice in one of four experimental arms: 1) Portfolio Plus diet and intensive increased physical activity program, 2) Portfolio Plus diet and a copy of Health Canada Physical Activity Guidelines with advice to increase physical activity, 3) DASH-like diet and an intensive increased physical activity program and 4) DASH-like diet and a copy of Health Canada Physical Activity Guidelines with advice to increase physical activity. The results of the study will have a major influence on dietary and exercise guidelines for coronary heart disease (CH risk reduction and provide evidence for the larger international trial that will focus on hard endpoints, myocardial infarction (MI) and CHD events). It is hoped that this cohort of participants will continue on and form part of the planned 9 year hard end point (MACE) study if funded.

Prior to starting treatments, participants will undergo screening ultrasound examination of both right and left carotids to enable selection of those individuals whose intima-media thickness (IMT) would be 5-30% below the cut point considered by the Mannheim Consensus as relevant arterial thickening to ensure a relatively low risk group, yet with some measurable arterial thickening.

It will be emphasized at the outset that both the dietary portfolio and the DASH-like diets have been associated with benefits in terms of cholesterol reduction to provide equal encouragement for all study arms. Portfolio and DASH-like dietary advice will consist of half hour individual sessions with the dietitian at baseline, and at 3-month intervals throughout the trial except for the first month when dietary advice will be reinforced, every 2 weeks, by telephone call to the participant or participant visit to the clinic. Prior to starting each diet, instruction will be given on achieving the dietary goals. At follow-up visits, the participants' completed 7-day diet records will be discussed and the original advice reinforced.

For the treatments with intensive increased physical activity the standardized physical activity/exercise component will be supervised by trained kinesiologists (exercise physiologists) for the 4 visits followed by monthly phone calls for the first year for the exercise component, when the major exercise training is provided. 7-day Exercise diaries will be collected at each visit. Using well-established procedures standardized across centers by the Quebec Heart and Lung Institute, the baseline visit will be used to provide a broad qualitative assessment of participants' lifestyle habits and preferences. Standardized physical activity questionnaires will be completed and participants will be asked to wear a pedometer for seven days prior to the intervention to quantify baseline physical activity (daily step count Cardiorespiratory fitness (CRF) is assessed using a submaximal treadmill test adapted from a progressive submaximal power output test performed on a cycle ergometer. The protocol begins with a warm-up workload of 2.5 mph with a 0% slope. The second stage is performed at a speed of 3.5 mph with a 2% slope. The third stage is adjusted in an attempt to reach 75% of the age-estimated maximal heart rate (HR). If necessary, a 4th stage is performed. Estimated VO2max is predicted by extrapolation to age-predicted maximal heart rate at a standardized submaximal treadmill stage (3.5 mph, 2% slope) and estimated maximal oxygen consumption (VO2max) are the variables considered as indicators of CRF in the present study.

For treatments with routine advice to increase physical activity, Health Canada Physical Activity Guidelines for adults 18-64 years or for older adults 65 years & older will be provided. They will be seen at the start and the end of each year for their formal exercise testing and will bring with them completed physical activities questionnaires. They will receive no other physical activities instruction.

Every effort will be made to obtain study blood samples and carotid imaging data from all subjects at the designated times regardless of adherence to the dietary aspects of the study protocol. All subjects will be included in the intention-to-treat analysis.

ELIGIBILITY:
A) Inclusion Criteria:

* Eligible participants will be

  * men over 21 years
  * post-menopausal women

Having a BMI less than or equal to 40 kg/m2 and who have measurable arterial thickening (>/=1.2mm) at screening as assessed by ultrasound.

They will include those who have at least 1 of the following characteristics:

1. Type 2 diabetes
2. Non-diabetic subjects post MI or post percutaneous coronary intervention (angioplasty) on statin therapy;
3. Hyper-cholesterolemic and treated with statins or have been prescribed statins but are not taking it because they are either unable (intolerant) or unwilling to take statin drugs.
4. Raised blood pressure, >140/90 (untreated)

B) Exclusion Criteria:

* Individuals with the following conditions will be excluded:

  * cardiovascular disease that precludes exercise e.g.

    * recent stroke or
    * recent myocardial infarction or
  * cardiac condition that severely compromises normal function:

    * mitral valve disease, atrial fibrillation and individuals with Implantable Cardioverter Defibrillator (ICD)
    * heart failure--grades 2-4 (based on New York Heart Association classification),
    * severe angina sufficient to prevent any form of physical activity
    * other conditions preventing exercise.
* secondary causes of hypercholesterolemia e.g. hypothyroidism (unless treated and on a stable dose of L-thyroxin), clinically significant renal (that precludes dietary change) or liver disease .
* LDL-cholesterol <1.4mmol/L
* uncontrolled blood pressure
* major disability
* disorder requiring continuous medical attention (on Coumadin) and treatment, such as:

  * chronic heart failure
  * liver disease
  * renal failure or
  * cancer (except non-melanoma skin cancer--basal cell, squamous cell)
  * chronic infections (bacterial or viral)
  * chronic inflammatory diseases (eg. lupus, ulcerative colitis, crohn's disease, celiac disease or gluten sensitivity)
  * other autoimmune disease
* major surgery <6 months prior to randomization
* newly diagnosed with diabetes (<3 months)
* alcohol consumption >3 drinks/d
* not suitable for MRI examination because of metal implants or claustrophobia
* food allergies or sensitivity to study foods or study food components (eg. tree nuts, peanuts, soy, wheat, gluten, oats, eggs, milk)
* already following a portfolio-like diet (and are not prepared to change) or have a structured exercise program which they cannot increase any further
* do not have a family doctor

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the maximum vessel wall volume of the carotid arteries by MRI at year 1 and 3 | At months 0, 12 and 36
  MRI imaging assessment of the carotid arteries will be done at baseline, end of year 1 and year 3.

SECONDARY OUTCOMES:
Coronary atheroma in the large vessels by MRI at year 1 and 3 | At months 0, 12 and 36
  This will be assessed by MRI imaging of the Coronary and carotid arteries
Lipid rich necrotic core by MRI at year 1 and 3 | At months 0, 12 and 36
  This will be assessed by MRI imaging of the Coronary and carotid arteries
intra plaque hemorrhage by MRI at year 1 and 3 | At months 0, 12 and 36
  This will be assessed by MRI imaging of the Coronary and carotid arteries
Blood pressure and pulse rate | At months 0, 12 and 36
  This is a composite measure that would by done using an automatic digital BP monitor which simultaneously measures and displays systolic and diastolic pressure (mmHg) and pulse rate (bpm) readings on an output screen.
Treatment difference in initiation of statin therapy | At month 12 and 36
  Assessment will be based on the current Canadian Cardiovascular Society Guidelines
Composite endpoint of Myocardial Infarction, Revascularization, Cardio Vascular hospitalization, Cardiovascular mortality and stroke | at month 12 and 36
  Information will be obtained from medical records of participants affected
Atrial Fibrillation and heart failure | at month 12 and 36
  Information will be obtained from medical records of the participants

OTHER OUTCOMES:
Completeness of clinic attendance and data collection and provision of fasting blood samples for planned tests. | At months -3, -0.5, and then at months 0, 3, 6, 9,12, 15, 18, 21, 24, 27, 30, 33 and 36
  This will be used as a measure of retention
Serum lipids: total cholesterol, LDL-chol, HDL-chol, and Triglycerides | At months -3, -0.5, and then at months 0, 3, 6, 9,12, 15, 18, 21, 24, 27, 30, 33 and 36
  Serum lipids will be measured at each Centre on fasting serum. LDL-C will be calculated using the Friedewald equation. Serum lipid standards will be used to quality control the lipid analyses at the collaborating sites
Hemoglobin A1c | At months -3, -0.5, 0, 3, 6, 9,12, 15, 18, 21, 24, 27, 30, 33 and 36
  safety monitoring especially for participants with type 2 diabetes
C-reactive protein | At months 0,12, 24 and 36
  C-reactive protein will be measured at each Centre on fasting serum.
Urinary analyses | At baseline (months -0.5 & 0) and end (months 33 & 36)
  24 hr urine samples will be analyzed for creatinine, urea, C-peptide, minerals, electrolytes and other dietary biomarkers
Fasting blood Glucose | At months -3, -0.5, 0, 3, 6, 9,12, 15, 18, 21, 24, 27, 30, 33 and 36
  safety monitoring especially for participants with type 2 diabetes
Blood Pressure | At months -3, -0.5, and then at months 0, 3, 6, 9,12, 15, 18, 21, 24, 27, 30, 33 and 36
  In clinic assessment using a digital blood pressure monitor
Treadmill testing | At month -1, and end of years 1, 2, and 3
  Physical fitness testing to assess fitness level
Diet history | At months -3, -0.5, and then at months 0, 3, 6, 9,12, 15, 18, 21, 24, 27, 30, 33 and 36
  7-day food records brought in at 3 monthly intervals will be analysed for macro and micro nutrient intakes.
Exercise history | At months -3, -0.5, and then at months 0, 3, 6, 9,12, 15, 18, 21, 24, 27, 30, 33 and 36
  7-day exercise/ activity records of the week prior to each study visit will be assessed for the type and duration of activity.
Pedometer records | At months -3, -0.5, and then at months 0, 3, 6, 9,12, 15, 18, 21, 24, 27, 30, 33 and 36
  These will be assessed for the daily step count over a 7-day period prior to the specified time points for the test group only.
Survey on quality of life | At months 0 and 36.
  This will be done using a Medical Outcomes Study 36-Item Short Form Questionnaire (SF-36).
Palatability (taste) of diet | At months 3, 6, 9,12, 15, 18, 21, 24, 27, 30, 33 and 36
  This will be measure on a scale to 1 to 10. 1 being 'strongly dislike' and 10 being 'like very much'. Participants will rate the taste (palatability) of the study diet and dietary components.
Satiety | At months 3, 6, 9,12, 15, 18, 21, 24, 27, 30, 33 and 36
  Using a 9-point bipolar semantic scale where -4 is extremely hungry, 0 is neutral and +4 is uncomfortably full, participants will rate their overall feeling of satiety for the previous week
Sustainability of diet (preparedness to continue on the diet) | At months 33 and 36
  Participants' preparedness to continue on the diet will be measured on a scale of 1 to 10. 1 = diet not sustainable; 10 = diet very sustainable
Genetic testing for specific genes | Week 0 or any other time point
  One time sample collection of buffy coat (from white cells) for future study on gene, diet, exercise and chronic disease relationship
Complete blood count (CBC) | Months 0, 12, 24 and 36
  Health check at start and yearly intervals
Renal function tests | Months 0, 12, 24 and 36
  Health check at start and yearly intervals
Liver function tests | Months 0, 12, 24 and 36
  Health check at start and yearly intervals
Prostatic specific antigen (PSA) | Months 0, 12, 24 and 36
  Health check at start and yearly intervals for male participants
Cognitive Assessment | months 0, 12, 24 and 36
  The Montreal Cognitive Assessment (MoCA) (version 7.1 original version) will be administered at months 0, 12, 24 and 36. This tool measures different cognitive domains such as attention, concentration, memory, language etc.

CONTACTS AND LOCATIONS:
Overall Officials: David Jenkins, MD, Principal Investigator — Risk Factor Modification Centre, St. Michael's Hospital; Benoit Lamarche, PhD, Study Director — Laval University; Peter Jones, PhD, Study Director — University of Manitoba; Jiri Frohlich, MD, Study Director — University of British Columbia
Locations (4):
- Canada (4):
  - Healthy Heart Lipid Clinic, St. Paul's Hospital, Vancouver, British Columbia
  - Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba, Winnipeg, Manitoba
  - Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario
  - Institute of Nutraceuticals and Functional Foods, Laval University, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Krauss RM, Eckel RH, Howard B, Appel LJ, Daniels SR, Deckelbaum RJ, Erdman JW Jr, Kris-Etherton P, Goldberg IJ, Kotchen TA, Lichtenstein AH, Mitch WE, Mullis R, Robinson K, Wylie-Rosett J, St Jeor S, Suttie J, Tribble DL, Bazzarre TL. AHA Dietary Guidelines: revision 2000: A statement for healthcare professionals from the Nutrition Committee of the American Heart Association. Circulation. 2000 Oct 31;102(18):2284-99. doi: 10.1161/01.cir.102.18.2284. No abstract available. PMID 11056107
- [Background] Anderson TJ, Gregoire J, Hegele RA, Couture P, Mancini GB, McPherson R, Francis GA, Poirier P, Lau DC, Grover S, Genest J Jr, Carpentier AC, Dufour R, Gupta M, Ward R, Leiter LA, Lonn E, Ng DS, Pearson GJ, Yates GM, Stone JA, Ur E. 2012 update of the Canadian Cardiovascular Society guidelines for the diagnosis and treatment of dyslipidemia for the prevention of cardiovascular disease in the adult. Can J Cardiol. 2013 Feb;29(2):151-67. doi: 10.1016/j.cjca.2012.11.032. PMID 23351925
- [Background] Ornish D, Scherwitz LW, Billings JH, Brown SE, Gould KL, Merritt TA, Sparler S, Armstrong WT, Ports TA, Kirkeeide RL, Hogeboom C, Brand RJ. Intensive lifestyle changes for reversal of coronary heart disease. JAMA. 1998 Dec 16;280(23):2001-7. doi: 10.1001/jama.280.23.2001. PMID 9863851
- [Background] Jenkins DJ, Chiavaroli L, Wong JM, Kendall C, Lewis GF, Vidgen E, Connelly PW, Leiter LA, Josse RG, Lamarche B. Adding monounsaturated fatty acids to a dietary portfolio of cholesterol-lowering foods in hypercholesterolemia. CMAJ. 2010 Dec 14;182(18):1961-7. doi: 10.1503/cmaj.092128. Epub 2010 Nov 1. PMID 21041432
- [Background] Jenkins DJ, Kendall CW, McKeown-Eyssen G, Josse RG, Silverberg J, Booth GL, Vidgen E, Josse AR, Nguyen TH, Corrigan S, Banach MS, Ares S, Mitchell S, Emam A, Augustin LS, Parker TL, Leiter LA. Effect of a low-glycemic index or a high-cereal fiber diet on type 2 diabetes: a randomized trial. JAMA. 2008 Dec 17;300(23):2742-53. doi: 10.1001/jama.2008.808. PMID 19088352
- [Background] Jenkins DJ, Kendall CW, Augustin LS, Mitchell S, Sahye-Pudaruth S, Blanco Mejia S, Chiavaroli L, Mirrahimi A, Ireland C, Bashyam B, Vidgen E, de Souza RJ, Sievenpiper JL, Coveney J, Leiter LA, Josse RG. Effect of legumes as part of a low glycemic index diet on glycemic control and cardiovascular risk factors in type 2 diabetes mellitus: a randomized controlled trial. Arch Intern Med. 2012 Nov 26;172(21):1653-60. doi: 10.1001/2013.jamainternmed.70. PMID 23089999
- [Background] Jenkins DJ, Kendall CW, Faulkner D, Vidgen E, Trautwein EA, Parker TL, Marchie A, Koumbridis G, Lapsley KG, Josse RG, Leiter LA, Connelly PW. A dietary portfolio approach to cholesterol reduction: combined effects of plant sterols, vegetable proteins, and viscous fibers in hypercholesterolemia. Metabolism. 2002 Dec;51(12):1596-604. doi: 10.1053/meta.2002.35578. PMID 12489074
- [Background] Borel AL, Nazare JA, Smith J, Almeras N, Tremblay A, Bergeron J, Poirier P, Despres JP. Visceral and not subcutaneous abdominal adiposity reduction drives the benefits of a 1-year lifestyle modification program. Obesity (Silver Spring). 2012 Jun;20(6):1223-33. doi: 10.1038/oby.2011.396. Epub 2012 Jan 19. PMID 22262155
- [Background] Borel AL, Nazare JA, Smith J, Almeras N, Tremblay A, Bergeron J, Poirier P, Despres JP. Improvement in insulin sensitivity following a 1-year lifestyle intervention program in viscerally obese men: contribution of abdominal adiposity. Metabolism. 2012 Feb;61(2):262-72. doi: 10.1016/j.metabol.2011.06.024. Epub 2011 Aug 23. PMID 21864868
- [Background] Pelletier-Beaumont E, Arsenault BJ, Almeras N, Bergeron J, Tremblay A, Poirier P, Despres JP. Normalization of visceral adiposity is required to normalize plasma apolipoprotein B levels in response to a healthy eating/physical activity lifestyle modification program in viscerally obese men. Atherosclerosis. 2012 Apr;221(2):577-82. doi: 10.1016/j.atherosclerosis.2012.01.023. Epub 2012 Jan 20. PMID 22321874
- [Background] Liu S, Willett WC, Stampfer MJ, Hu FB, Franz M, Sampson L, Hennekens CH, Manson JE. A prospective study of dietary glycemic load, carbohydrate intake, and risk of coronary heart disease in US women. Am J Clin Nutr. 2000 Jun;71(6):1455-61. doi: 10.1093/ajcn/71.6.1455. PMID 10837285
- [Background] Pereira MA, O'Reilly E, Augustsson K, Fraser GE, Goldbourt U, Heitmann BL, Hallmans G, Knekt P, Liu S, Pietinen P, Spiegelman D, Stevens J, Virtamo J, Willett WC, Ascherio A. Dietary fiber and risk of coronary heart disease: a pooled analysis of cohort studies. Arch Intern Med. 2004 Feb 23;164(4):370-6. doi: 10.1001/archinte.164.4.370. PMID 14980987
- [Background] Keys A, Aravanis C, Blackburn HW, Van Buchem FS, Buzina R, Djordjevic BD, Dontas AS, Fidanza F, Karvonen MJ, Kimura N, Lekos D, Monti M, Puddu V, Taylor HL. Epidemiological studies related to coronary heart disease: characteristics of men aged 40-59 in seven countries. Acta Med Scand Suppl. 1966;460:1-392. No abstract available. PMID 5226858
- [Background] Shai I, Schwarzfuchs D, Henkin Y, Shahar DR, Witkow S, Greenberg I, Golan R, Fraser D, Bolotin A, Vardi H, Tangi-Rozental O, Zuk-Ramot R, Sarusi B, Brickner D, Schwartz Z, Sheiner E, Marko R, Katorza E, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Stampfer MJ; Dietary Intervention Randomized Controlled Trial (DIRECT) Group. Weight loss with a low-carbohydrate, Mediterranean, or low-fat diet. N Engl J Med. 2008 Jul 17;359(3):229-41. doi: 10.1056/NEJMoa0708681. PMID 18635428
- [Background] Touboul PJ, Hennerici MG, Meairs S, Adams H, Amarenco P, Desvarieux M, Ebrahim S, Fatar M, Hernandez Hernandez R, Kownator S, Prati P, Rundek T, Taylor A, Bornstein N, Csiba L, Vicaut E, Woo KS, Zannad F; Advisory Board of the 3rd Watching the Risk Symposium 2004, 13th European Stroke Conference. Mannheim intima-media thickness consensus. Cerebrovasc Dis. 2004;18(4):346-9. doi: 10.1159/000081812. Epub 2004 Nov 2. PMID 15523176
- [Background] Jenkins DJ, Kendall CW, Faulkner DA, Nguyen T, Kemp T, Marchie A, Wong JM, de Souza R, Emam A, Vidgen E, Trautwein EA, Lapsley KG, Holmes C, Josse RG, Leiter LA, Connelly PW, Singer W. Assessment of the longer-term effects of a dietary portfolio of cholesterol-lowering foods in hypercholesterolemia. Am J Clin Nutr. 2006 Mar;83(3):582-91. doi: 10.1093/ajcn.83.3.582. PMID 16522904
- [Background] The DASH diet. Dietary Approaches to Stop Hypertension. Lippincotts Prim Care Pract. 1998 Sep-Oct;2(5):536-8. No abstract available. PMID 9791393
- [Background] Murie-Fernandez M, Irimia P, Toledo E, Martinez-Vila E, Buil-Cosiales P, Serrano-Martinez M, Ruiz-Gutierrez V, Ros E, Estruch R, Martinez-Gonzalez MA; PREDIMED Investigators. Carotid intima-media thickness changes with Mediterranean diet: a randomized trial (PREDIMED-Navarra). Atherosclerosis. 2011 Nov;219(1):158-62. doi: 10.1016/j.atherosclerosis.2011.06.050. Epub 2011 Jul 6. PMID 21802081
- [Derived] Kavanagh ME, Chiavaroli L, Quibrantar SM, Viscardi G, Ramboanga K, Amlin N, Paquette M, Sahye-Pudaruth S, Patel D, Grant SM, Glenn AJ, Ayoub-Charette S, Zurbau A, Josse RG, Malik VS, Kendall CWC, Jenkins DJA, Sievenpiper JL. Acceptability of a Web-Based Health App (PortfolioDiet.app) to Translate a Nutrition Therapy for Cardiovascular Disease in High-Risk Adults: Mixed Methods Randomized Ancillary Pilot Study. JMIR Cardio. 2025 Mar 28;9:e58124. doi: 10.2196/58124. PMID 40152922

DOCUMENTS (1):
  • Study Protocol (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT02481466/Prot_000.pdf